CLINICAL TRIAL: NCT05210400
Title: Prospectively Assessing Pain After Breast Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Scott Karlan, M.D., Cedars-Sinai Medical Center
Other Study IDs: STUDY00001859
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Reducing post-operative pain and reducing the use of opioid narcotics are independently valuable goals. Before studying newer techniques that may help us achieve these goals, we need objective data on how much pain normally occurs after breast surgery done with standard-of-care techniques. This study was designed to obtain baseline data.

DETAILED DESCRIPTION:
Breast surgeons may be able to reduce post-operative pain and the need for opioid narcotics by utilizing regional anesthesia techniques (modified regional blocks) during surgery. To test this hypothesis, we need baseline (pre-intervention) data on how much pain patients experience when breast surgery is done without blocks.

In this study, we will gather data on (1.) pain pills used after surgery, and (2.) pain scores in the recovery room. This will allow us to establish how much pain normally occurs after axillary surgery (sentinel node biopsy or axillary dissection), with or without concurrent lumpectomy, done by a participating breast surgeon.

After analyzing this data, our plan is to do a second study, with a new group of patients, to assess whether there is any change in outcome after surgeons implement these new techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Female, age 18 or older.
4. Scheduled for axillary surgery (sentinel node biopsy or axillary dissection), with or without concurrent lumpectomy.
5. Able to take oral narcotics and be willing to adhere to the prescribed regimen.

Exclusion Criteria:

1. A history of chronic pain
2. Any previously diagnosed chronic pain syndrome.
3. Prior use of narcotics, on more than 5 days in the past 3 months or 10 days in the past year.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Recruitment will depend on referral by one of the study co-investigators, at the time that they schedule a patient for axillary surgery with or without concurrent lumpectomy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Pain scores in recovery room | The day of surgery
  EMR documentation from the recovery room
Number of narcotic pain pills used after surgery | Assessed approximately a week after surgery